CLINICAL TRIAL: NCT04229407
Title: A Post-marketing, Double-blind, Placebo-controlled, Randomized, Parallel Study to Evaluate the Effect of Dietary Supplement on Muscle Mass and Physical Performance Among People Aged 50 Years and Older
Brief Title: Evaluate the Effect of Dietary Supplement on Muscle Mass and Physical Performance for Over 50 Years Old People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Orient Europharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OEP-6CR003-401
Record Dates: First submitted 2018-04-10; First posted 2020-01-18 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Muscle Loss
MeSH Terms: conditions — Muscular Atrophy | interventions — Dietary Supplements; Folic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary supplement (Experimental): subject will be evaluated for the eligibility of MRI assessment to assign subjects in randomization strata (MRI or non-MRI).
  After 32 subjects in MRI strata is reached. subjects will be randomized to intake Dietary supplement twice daily (every morning and night, 30 minutes after exercise if do exercise) for 12 weeks
  Interventions: Dietary Supplement: Dietary supplement
- vitamin B (Placebo Comparator): subject will be evaluated for the eligibility of MRI assessment to assign subjects in randomization strata (MRI or non-MRI).
  After 32 subjects in MRI strata is reached. subjects will be randomized to intake placebo vitamin B twice daily (every morning and night, 30 minutes after exercise if do exercise) for 12 weeks.
  Interventions: Dietary Supplement: vitamin B

INTERVENTIONS:
Dietary Supplement: Dietary supplement — MRI eligibility evaluation Dietary supplement drink powder dissolved in 150 c.c. warm water oral intake twice daily at every morning and night (30 minutes after exercise if do exercise) for 12 weeks subjects will be instructed to do 45-minute exercise once a week following the training program of the study trainer at gym, and 30-minute exercise (per exercise manual) at least twice a week at home.
  Arms: Dietary supplement
Dietary Supplement: vitamin B — MRI eligibility evaluation vitamin B drink powder dissolved in 150 c.c. warm water oral intake twice daily at every morning and night (30 minutes after exercise if do exercise)for 12 weeks subjects will be instructed to do 45-minute exercise once a week following the training program of the study trainer at gym, and 30-minute exercise (per exercise manual) at least twice a week at home.
  Arms: vitamin B

SUMMARY:
To assess the ability and safety profile of dietary supplement to augment lean body mass, muscle strength, and physical performance among people aged 50 years and older

DETAILED DESCRIPTION:
In light of the rapidly expanding aging population, sarcopenia and related disorders are emerging as a major public health problem of the 21st century.Sponsor has produced a dietary supplement, which has been on market in Taiwan. The proposed study is conducted to confirm whether the amino acid supplementation is able to enhance the magnitude of gain in lean body mass and muscle strength in middle-aged and older adults with muscle loss or sarcopenia undergoing exercise training.

ELIGIBILITY:
Main Inclusion Criteria:

1. Male or female aged 50 years or older.
2. Subjects who has muscle loss or at risk of muscle loss, with symptoms of reduced physical activities, reduced gait speed, exhaustion, or had tumbled/ fallen within past year
3. Willing to comply with study procedures and follow-ups
4. Provide written consent

Main Exclusion Criteria:

1. Gait speed ≤ 0.3 m/sec
2. Any disease that interferes with limb function, including:

   1. Limb fracture within past 6 months
   2. Severe knee, hip, or arm arthritis
   3. As judged by the investigator, disorder of nervous system (i.e., stroke, severe spinal stenosis, peripheral neuropathy, and Parkinson's disease) with poor control
   4. Intermittent claudication due to peripheral artery disease
3. As judged by the investigator, mental disorders (i.e., confirmed diagnosis of dementia) with poor control
4. Cardiopulmonary disease with poor control judged by the investigator
5. Malignancy with poor control judged by the investigator
6. Subjects claim to have chronic renal disease, defined as kidney damage or GFR < 30 mL/min/1.73 m2 for at least 3 months
7. Severe visual and hearing impairment that becomes barrier to communication
8. Subjects have taken any hormone replacement therapy within 3 months prior to study enrollment, or plans to begin hormone replacement therapy at any time during the study
9. Subjects with known poorly controlled diabetes (HbA1c > 9.0%), hyperthyroidism or thyroid insufficiency, Cushing's syndrome, or adrenal insufficiency
10. Subjects with known milk allergy or lactose intolerance
11. Other conditions that investigator considers subject is ineligible to participate in the study

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2020-10-07 (Actual); Study Completion 2020-10-07 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects achieving clinically meaningful improvement in Increment ≥ 3% in bone-free lean body mass (unit: kilogram) at 12 weeks after baseline | 12 weeks
  Bone-free lean body mass will be assessed by measured by dual- energy X-ray absorptiometry. An increment of ≥ 3% from baseline after 12 weeks of intervention will be regarded as clinically meaningful improvement.
The proportion of subjects achieving clinically meaningful improvement in Increment ≥ 3% in 30-sec chair stand test (unit: number of stand) at 12 weeks after baseline | 12 weeks
  The score is the total number of stands within 30 seconds.
The proportion of subjects achieving clinically meaningful improvement in Increment ≥ 3% in strength of hand grip (unit: kilogram) at 12 weeks after baseline | 12 weeks
  Strength of hand grip will be assessed by Smedlay's DynamoMeter TTM Tokyo Japan. An increment of ≥ 3% from baseline after 12 weeks of intervention will be regarded as clinically meaningful improvement.

SECONDARY OUTCOMES:
Mean change in bone-free lean body mass at 4 and 12 weeks after baseline | 12 weeks
  Bone-free lean body mass will be assessed by measured by dual- energy X-ray absorptiometry.
Mean change in 30-sec chair stand test at 4 and 12 weeks after baseline | 12 weeks
  The score is the total number of stands within 30 seconds.
Mean change in 6-meter walk test at 4 and 12 weeks after baseline | 12 weeks
  The 6MWT measures the walking speed an individual is able to walk over a total of six meters on a hard, flat surface at their usual pace.
Mean change in short physical performance battery (SPPB) score at 4 and 12 weeks after baseline | 12 weeks
  including Balance test, Gait speed test, Chair stand test
Mean change in strength of hand grip at 4 and 12 weeks after baseline | 12 weeks
  Strength of hand grip will be assessed by Smedlay's DynamoMeter TTM Tokyo Japan.
Mean change in intramuscular fat assessed by MRI at 12 weeks after baseline | 12 weeks
  Intramuscular fat will be assessed using the magnetic resonance images (MRI) at baseline and Week 12 for 32 subjects.
Adverse events | 12 weeks
  Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Liang-Kung Chen, MD.PhD, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Veteran General Hospital-Taipei, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No